CLINICAL TRIAL: NCT03630666
Title: A Study Comparing Intermittent Androgen Depriving Therapy With Or Without Salvage High-Dose Intensity Modulation Radiotherapy (IG-IMRT)To Oligometastatic Pelvic Lymph Nodes In Biochemically-relapsing Prostate Cancer Patients.
Brief Title: Comparison of Intermittent Androgen Deprivation Therapy With or Without Irradiation Recovery in Prostate Cancer Patients
Acronym: OLIGOPELVIS2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2017-13
Record Dates: First submitted 2018-07-04; First posted 2018-08-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Oligometastasis
Keywords: Oligometastatic pelvic lymph nod, IADT, radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Radiotherapy

STUDY DESIGN:
Intervention Model Description: phase 3 study, randomised, open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IADT - Intermittent Androgen Deprivation Therapy (Active Comparator): one injection of IADT. The overall duration of IADT will be six months.
  Interventions: Drug: IADT
- IADT + Radiotherapy (Intermittent Androgen Deprivation Therapy plus Radiotherapy) (Experimental): One injection of IADT. The overall duration of IADT will be six months. Irradiation three months after injection of IADT. The overall duration of radiotherapy will be three months.
  Interventions: Combination Product: IADT + radiotherapy

INTERVENTIONS:
Drug: IADT — Patient will receive one injection of IADT at randomization
  Other Names: LH-RH (Luteinizing Hormone Releasing Hormone) agonist
  Arms: IADT - Intermittent Androgen Deprivation Therapy
Combination Product: IADT + radiotherapy — Patient will receive one injection of IADT at randomization then will receive irradiation 3 months after injection of IADT
  Other Names: IG-IMRT; LH-RH (Luteinizing Hormone Releasing Hormone) agonist
  Arms: IADT + Radiotherapy (Intermittent Androgen Deprivation Therapy plus Radiotherapy)

SUMMARY:
Metastatic prostate cancer has traditionally been regarded as an incurable dissemination of disease, and treatment is focused on delaying progression rather than eliminating all tumor burden. Local therapies, and specifically radiotherapy, have been directed at quality of life endpoints and not at improving survival. However, advances in imaging and systemic therapy have identified a population of 'oligometastatic' patients who have a lower burden of metastatic disease (usually ≤5 lesions), who may present an exception. This condition is hypothesized to occupy the hinterland between incurable metastatic disease and locoregional disease, where micrometastatic disease is assumed to exist and yet remain eradicable. Oligometastases can be detected using standard imaging but the sensitivity of these exams is very low for patients with a PSA below 10 ng/ml. In France, FCH PET imaging is now routinely available in a large majority of cancer centres. More recently, PSMA PET imaging has been developed.

Since most oligometastases are now discovered at a time when conventional imaging is unable to detect metastases, we must rely on the literature regarding purely biochemically-relapsing prostate cancer patients. Three strategies have been explored: (i) observation until symptoms develop, (ii) early intermittent Androgen Deprivation Therapy (IADT) and (iii) continuous Androgen Deprivation Therapy (ADT). Recent data suggest that, of the three strategies, early intermittent ADT was superior in term of overall survival to observation in controlling metastatic prostate cancer, and this effect was similar in the biochemically-relapsing prostate cancer patient population.

This phase III study will explore the role of salvage pelvic IG-IMRT combined with intermittent ADT (IADT) in pelvic oligometastatic patients in prolonging the first failure-free interval between the first and the second intermittent ADT courses.

DETAILED DESCRIPTION:
Screening procedures will be performed up to three months before starting IADT. After obtaining informed consent, patients will be randomly allocated to one of two groups:

Experimental group: IADT + IG-IMRT Control group: IADT

In both study arms, the first injection of IADT will be administered in hospital on the day of randomization. The overall duration of IADT will be six months.

In the experimental group, patients will receive radiotherapy three months after the first injection of IADT.

The overall duration of radiotherapy will be three months.

The overall duration of IADT will be six months. It will be administered three months, +/- 15 days prior to the first day of radiotherapy. At the completion of the six-month treatment period, a non-treatment interval will start if :

there is no evidence of clinical disease progression and the PSA level is ≤ 4.00 ng/ml If the PSA subsequently rises above 0.20 ng/ml and is confirmed by a second measurement at least three weeks later, PET/CT imaging will be repeated every 6 months until a clinical failure is detected or until the PSA rises above 4.00 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven prostate adenocarcinoma
* Age ≥ 18 years
* Performance Status 0-1
* Prior radical prostate treatment (surgery and/or radiotherapy)
* ≤ 5 metastatic pelvic lymph nodes detected by FCH-PET or PSMA-PET
* Upper limit of metastatic lymph nodes: aortic bifurcation
* If ADT has been previously administered to the patient, at least 12 months must have elapsed between the predicted duration of the last injection and inclusion of the patient in the study. For this category of patients, serum testosterone must be higher than 6 nmol/L (50 ng/L) prior to inclusion
* Biochemical relapse (according to the European Association of Urology guidelines) is defined by :

Following radical prostatectomy (RP), biochemical recurrence (BCR) is defined by two consecutive rising PSA values > 0.20 ng/ml After primary radiation therapy (RT), the Radiation Therapy Oncology Group (RTOG) and American Society for Radiation Oncology Phoenix Consensus Conference definition of PSA failure is any PSA increase > 2.00 ng/ml higher than the PSA nadir value, regardless of the serum concentration of the nadir.

* Having given written informed consent prior to any procedure related to the study.
* Patient is willing and able to comply with the protocol for the duration of the study including all scheduled treatment, visits and examinations.
* Patient has valid health insurance
* Subjects who have partners of childbearing potential must be willing to use a method of effective birth control during treatment and for 12 months following completion of treatment with ADT or IG-IMRT.

Exclusion Criteria:

* Bone or visceral metastases
* Para-aortic lymph node metastases (above the aortic bifurcation)
* Presence of more than five metastatic lymph nodes
* Evidence of local intra-prostatic relapse
* Evidence of prostate bed relapse in a previously irradiated region. Prostate bed relapses which have not been previously irradiated will not be excluded
* Evidence of metastasis at initial diagnosis
* Evidence of distant metastases beyond the pelvic lymph nodes
* Previous irradiation of pelvic lymph nodes
* Castration-resistant prostate cancer (CRPC) as defined by : a castrate serum testosterone < 6 nmol/L (50 ng/L)
* Contraindications to pelvic irradiation (e.g. chronic inflammatory bowel disease)
* Contraindications to ADT (known hypersensitivity to any of the study drugs or excipients)
* Severe uncontrolled hypertension defined as systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy
* Other malignancy treated within the last 5 years (except non-melanoma skin cancer)
* Patients with a biochemical relapse while on active treatment with LHRH-agonist, LHRH-antagonist, anti-androgen, maximal androgen blockade, or oestrogen
* Treatment during the past month with products known to influence PSA levels (such as finasteride)
* In case of previous prostate/prostate bed radiotherapy, PET-positive lymph nodes have to be located outside the previous irradiation field with a maximum of 20 Gy to the PET-positive lymph nodes region
* Patients already included in another therapeutic trial with an experimental drug or having been given an experimental drug within a period of 30 days
* Disorder precluding understanding of trial information or informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 90 months
  PSA or CT scan

SECONDARY OUTCOMES:
overall survival | 90 months
  death
time to castration-resistance | 90 months
  serum testosterone mesure
toxicity to IADT and radiation | 90 months
  evaluation with NCI-CTC AE v4.03
Quality of life during long-term treatment | Up to 90 months after start of treatment
  Quality of life will be assessed every 3 months using the EORTC QLQ-C30 and the prostate cancer-specific module QLQ-PR25. These validated questionnaires evaluate physical, emotional, and social functioning, as well as symptoms related to prostate cancer and its treatment.
site of tumor progression | 90 months
  FCH or PSMA PET at biochemical relapse

CONTACTS AND LOCATIONS:
Overall Officials: STEPHANE SUPIOT, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (16):
- France (16):
  - Institut Sainte Catherine, Avignon
  - Institut Bergonie, Bordeaux
  - CHRU de Brest, Brest
  - Clinique Pasteur, Brest
  - Institut de Cancérologie de Bourgogne, Chalon-sur-Saône
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut de Cancérologie de Montpellier, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Institut de Cancérologie, Nantes
  - Hopital Privé du Confluent, Nantes
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - ICL Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Saint Yves, Vannes